CLINICAL TRIAL: NCT06341010
Title: The Role of Angiojet Rheolytic Thrombectomy in The Management of Iliofemoral Deep Venous Thrombosis
Status: Recruiting | Type: Observational
Sponsor: Abdelrahman Ibrahim Sayed Mohamed Abdalla (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Ibrahim Sayed Mohamed Abdalla, faculty of medicine Assiut university, Assiut University
Organization: Assiut University (Other)
Other Study IDs: The Role of Angiojet Rheolytic
Record Dates: First submitted 2023-09-24; First posted 2024-04-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Iliofemoral Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Angiojet Rheolytic Thrombectomy in The Management of Iliofemoral Deep Venous Thrombosis — Angiojet Rheolytic Thrombectomy in The Management of Iliofemoral Deep Venous Thrombosis

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of rheolytic thrombectomy in restoring venous patency DVT, periprocedural complications and development of PTS after tratment of iliofemoral DVT.

DETAILED DESCRIPTION:
Deep venous thrombosis (DVT) is a common disease affecting approximately 0.1% of the world population.1 The incidence of DVT steadily increases as the patient gets older. One-third of patients with DVT may develop pulmonary embolism (PE)2. DVT can significantly influence the quality of life of patients, and it represents an important clinical and economic disease burden on health-care systems.

Over the years, different options for DVT treatment have been introduced to restore patency, save valve function, and reduce the occurrence of post-thrombotic syndrome (PTS).

The conventional treatment of acute DVT aims to prevent thrombus propagation and to reduce the risks of PE and DVT recurrence5. However, this treatment is ineffective at reducing thrombus burden and consequently does not prevent PTS. Recent advances in catheter-based interventions have led to the development of a variety of minimally invasive endovascular strategies to remove venous thrombus.

Lower-extremity DVT, especially proximal or iliofemoral DVT, has been demonstrated to confer the greatest risk for complications such as pulmonary embolism, thrombosis recurrence, and post- thrombotic syndrome. Most practice guidelines recommend early clot removal for patients with iliofemoral DVT who have symptoms less than 14 days in duration, good functional ability, and acceptable life expectancy and who are at low risk for bleeding complications.

Removal of clot can be achieved by using catheter-directed thrombolysis (CDT) or pharmacomechanical.Use of CDT is limited because of the lengthy procedure/hospitalization time and intensive care unit (ICU) stays required for the procedure11. pharmacomechanical was developed to address the limitations of CDT by combining catheter-based and mechanical technology to fragment and/or aspirate thrombus in addition to delivering a thrombolytic drug throughout the thrombus.

Percutaneous rheolytic thrombectomy (RT) technique is highly effective at clearing thrombus, which preserves venous valve function and prevents subsequent PTS. The use of RT to treat DVT may reduce long-term morbidity in DVT patients by restoring the patency of the veins and preventing pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

Acute IF DVT

life expectancy more than 1 year

Exclusion Criteria:

* Recurrence of DVT Chronic DVT The catheter cannot be used in vessels smaller than 6mm. Patients have contraindications for endovascular procedures Patients cannot tolerate contrast media In patients with lesions that cannot be accessed with the guide wire Pregnancy History of pelvic surgery with left iliac vein injury or pelvic radioactive therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients presented with acute iliofemoral DVT
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | Immediately intraoperative
  Thrombus removal and restoration of the venous flow intraoperatively

SECONDARY OUTCOMES:
Incidence of PTS | Two years
  Incidence of post-thrombotic syndrome within 2 years after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Asyut university, Asyut, Egypt

REFERENCES:
- [Background] Meissner MH, Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Lohr JM, McLafferty RB, Murad MH, Padberg F, Pappas P, Raffetto JD, Wakefield TW; Society for Vascular Surgery; American Venous Forum. Early thrombus removal strategies for acute deep venous thrombosis: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2012 May;55(5):1449-62. doi: 10.1016/j.jvs.2011.12.081. Epub 2012 Apr 1. PMID 22469503
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Dumantepe M, Uyar I. The effect of Angiojet rheolytic thrombectomy in the endovascular treatment of lower extremity deep venous thrombosis. Phlebology. 2018 Jul;33(6):388-396. doi: 10.1177/0268355517711792. Epub 2017 May 22. PMID 28530488